CLINICAL TRIAL: NCT01296724
Title: PREMAPIV : Intravesical Pressure Variation at Different Bladder Instillation Volumes in Newborn Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 2010-A01346-33; LOC/10-17
Record Dates: First submitted 2011-02-14; First posted 2011-02-15 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2013-11

CONDITIONS: Intensive Care Unit Syndrome

ARMS (2):
- newborn with digestive pathology (Other): Preterm or term newborn admitted in paediatric intensive care unit with an urethral catheter and digestive pathology
  Interventions: Other: Measure of intravesical pressure
- Newborn without digestive pathology (Other): Preterm or term newborn admitted in paediatric intensive care unit with an urethral catheter and without digestive pathology
  Interventions: Other: Measure of intravesical pressure

INTERVENTIONS:
Other: Measure of intravesical pressure — For the installation of the urinary catheter, a valve connected to a pressure head is intercalated between the probe and the collecting bag. Various Intravesical pressure measurements will be conducted after injection of 0 ml/kg, 0.5 ml/kg, 1 ml/kg, 1.5 ml/kg, 2 ml/kg, 2.5 ml/kg 3 ml/kg, 3.5 ml/kg and 4 ml/kg of physiological saline.
  Arms: newborn with digestive pathology
Other: Measure of intravesical pressure — For the installation of the urinary catheter, a valve connected to a pressure head is intercalated between the probe and the collecting bag. Various IVP measurements will be conducted after injection of 0 ml/kg, 0.5 ml/kg, 1 ml/kg, 1.5 ml/kg, 2 ml/kg, 2.5 ml/kg 3 ml/kg, 3.5 ml/kg and 4 ml/kg of physiological saline.
  Arms: Newborn without digestive pathology

SUMMARY:
Abdominal Compartment Syndrome (ASC) is defined by an Intra Abdominal Hypertension (IAH) associated with a new organ failure. The occurrence of this syndrome is not well known in infants. Preterm birth is frequently associated with gastrointestinal complications, particularly Necrotizing Enterocolitis. In this pathology it is likely that the intra abdominal pressure (IAP) increases and can participate in the occurrence of organ failures. Newborn, in particular with digestive malformation as diaphragmatic hernias, gastroschisis, could themselves be suffering from this syndrome. It would be interesting to make early diagnosis in order to optimize the management of these children. This requires reliable measurements methods and standards. Intravesical Pressure (IVP) is the most reliable validated indirect method to measure intra-abdominal pressure. In order to measure the IVP, the bladder must contain a minimum of liquid. However, using inappropriate volumes could give erroneous IAP readings. The optimal amount of saline to inject in older children, determined from pressure-volume curves study is 1 ml/kg. In preterm and term infants, this volume appear extremely low (e.g. 0 8cc if taking a child to 800 g). The question that arises is whether this quantity is sufficient to obtain reliable and reproducible measurements of IVP in preterm and term.

ELIGIBILITY:
Inclusion Criteria:

* Preterm or term newborn admitted in paediatric intensive care unit
* With an urethral catheter
* Consent signed by parents

Exclusion Criteria:

* Weight > 4.5 kg
* Urinary tract or bladder pathology

Max Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2011-02; Primary Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Determinate the optimal volume of saline injection in the bladder for measuring intravesical pressure in infants, with and without digestive pathology | 2 years

SECONDARY OUTCOMES:
Determine the normal intravesical pressure in critically ill children, with and without digestive pathology | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Tirel, Principal Investigator — Rennes University Hospital
Locations (1):
- Rennes University Hospital, Rennes, Brittany Region, France